CLINICAL TRIAL: NCT02738203
Title: Self-Administered Lidocaine Gel for Pain Management With IUD Insertion: A Randomized Controlled Trial
Brief Title: Self-Administered Lidocaine Gel for Pain Management With IUD Insertion
Acronym: SALUD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Conti, Clinical Instructor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32825
Record Dates: First submitted 2016-04-04; First posted 2016-04-14 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: IUD Insertion
Keywords: Pain Management; IUD insertion
MeSH Terms: conditions — Agnosia | interventions — Lidocaine; K-Y jelly

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental, IUD Insertion group (Experimental): If the subject is assigned to the experimental group (vaginal lidocaine jelly):
  She will be given a pre-filled vaginal inserter with 10 ml of 2% lidocaine jelly) and will be asked to insert it vaginally 20-30 minutes prior to the start of her procedure. The subject will not know if she received the active drug or a placebo.
  Interventions: Drug: Vaginal 2% Lidocaine
- Control, IUD Insertion group (Placebo Comparator): If the subject is assigned to the control group (sterile, surgical lubricant jelly):
  •She will be given a pre-filled vaginal inserter with 10 ml of surgical lubricant jelly and will be asked to insert it vaginally 20-30 minutes prior to the start of her procedure. The subject will not know if she received the active drug or a placebo.
  Interventions: Drug: Surgical Lubricant Jelly

INTERVENTIONS:
Drug: Vaginal 2% Lidocaine — Patient-administered vaginal Lidocaine jelly verse surgical lubricant jelly
  Arms: Experimental, IUD Insertion group
Drug: Surgical Lubricant Jelly — Patient-administered vaginal surgical lubricant jelly verse Lidocaine jelly
  Other Names: K-Y Jelly
  Arms: Control, IUD Insertion group

SUMMARY:
For intrauterine device (IUD) insertion, currently there are no standardized clinical guidelines for pain management. The investigators aim to explore whether adequate pain relief is possible through self-administered, non-invasive means alone. Reducing pain associated with IUD insertion may benefit patients and providers. When patients are comfortable during their procedure, it is likely the provider can more quickly and with fewer complications perform the insertion. The investigators propose to explore the effect of a locally applied vaginal lidocaine gel in place of the standard of care pain management, no intervention, prior to IUD insertions. This is a superiority, blinded, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

Elective IUD insertion (any type of IUD, copper or hormonal); at an out-patient setting at Stanford; English or Spanish speaking, and ability to give informed consent.

Exclusion Criteria:

Any pre-operative use of misoprostol; or use of PO pain control medication (i.e. ibuprofen or acetaminophen) prior to procedure. Allergy to study medications: lidocaine, or surgical lubricant jelly, known uterine anomaly; prior cervical surgery; and no prior use of tampons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Conti, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Gynecology Clinic, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conti JA, Lerma K, Schneyer RJ, Hastings CV, Blumenthal PD, Shaw KA. Self-administered vaginal lidocaine gel for pain management with intrauterine device insertion: a blinded, randomized controlled trial. Am J Obstet Gynecol. 2019 Feb;220(2):177.e1-177.e7. doi: 10.1016/j.ajog.2018.11.1085. Epub 2018 Nov 13. PMID 30444982

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental, IUD Insertion Group: If the subject is assigned to the experimental group (vaginal lidocaine jelly):
  She will be given a pre-filled vaginal inserter with 10 ml of 2% lidocaine jelly) and will be asked to insert it vaginally 20-30 minutes prior to the start of her procedure. The subject will not know if she received the active drug or a placebo.
  Vaginal 2% Lidocaine: Patient-administered vaginal Lidocaine jelly verse surgical lubricant jelly
- Control, IUD Insertion Group: If the subject is assigned to the control group (sterile, surgical lubricant jelly):
  •She will be given a pre-filled vaginal inserter with 10 ml of surgical lubricant jelly and will be asked to insert it vaginally 20-30 minutes prior to the start of her procedure. The subject will not know if she received the active drug or a placebo.
  Surgical Lubricant Jelly: Patient-administered vaginal surgical lubricant jelly verse Lidocaine jelly
Period: Overall Study
Arm/Group | Experimental, IUD Insertion Group | Control, IUD Insertion Group
Started | 110 | 110
Completed | 108 | 107
Not Completed | 2 | 3
Not completed — Failed IUD Insertion | 2 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Per protocol analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental, IUD Insertion Group | Control, IUD Insertion Group | Total
Number analyzed (Participants) | 108 | 107 | 215
Age, Continuous [Median (Full Range); unit: years] | 28.9 [18 to 48] | 27 [18 to 51] | 28 [18 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 107 | 215
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 15 | 29
  Not Hispanic or Latino | 93 | 90 | 183
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 14 | 17 | 31
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 5 | 5 | 10
  White | 69 | 67 | 136
  More than one race | 9 | 6 | 15
  Unknown or Not Reported | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 108 | 107 | 215
Previous Intrauterine Device Insertion [Count of Participants; unit: Participants] — Participant had a previous intrauterine device insertion.
  Participants | 37 | 33 | 70

OUTCOME MEASURES:

1. Primary Outcome: (IUD Insertion): Pain Perceived by Visual Analogue Scale (0-100 mm) Immediately Following Procedure Completion
Description: Pain immediately after speculum removal as measured by a Visual Analog Scale (VAS). This scale is 0-100--on the scale "0" had "no pain" and "100" had "worst pain imaginable" as anchors. A higher score indicates higher pain.
Time Frame: 0-3 minutes after procedure completed
Population: Per protocol analysis
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Experimental, IUD Insertion Group | Control, IUD Insertion Group
Number analyzed (Participants) | 108 | 107
score on a scale | 65 [1 to 99] | 59 [5 to 100]

2. Secondary Outcome: Anticipated Pain as Measured by a Visual Analog Scale
Description: Pain as measured by a Visual Analog Scale (VAS). This scale is 0-100--on the scale "0" had "no pain" and "100" had "worst pain imaginable" as anchors. A higher score indicates higher pain.
Time Frame: 30 Minutes prior to procedure
Population: Per protocol analysis
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Experimental, IUD Insertion Group | Control, IUD Insertion Group
Number analyzed (Participants) | 108 | 107
score on a scale | 60 [1 to 87] | 59 [6 to 94]

3. Secondary Outcome: Baseline Pain as Measured by a Visual Analog Scale
Description: as for outcome 2
Time Frame: Immediately prior to procedure; upon arrival to procedure room
Population: Per protocol analysis
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Experimental, IUD Insertion Group | Control, IUD Insertion Group
Number analyzed (Participants) | 108 | 107
score on a scale | 2 [0 to 77] | 2 [0 to 22]

4. Secondary Outcome: Pain After Speculum Placement as Measured by a Visual Analog Scale
Description: as for outcome 2
Time Frame: Intraoperative
Population: Per protocol analysis
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Experimental, IUD Insertion Group | Control, IUD Insertion Group
Number analyzed (Participants) | 108 | 107
score on a scale | 7 [0 to 81] | 11 [0 to 80]

5. Secondary Outcome: Pain After Tenaculum Placement as Measured by a Visual Analog Scale
Description: as for outcome 2
Time Frame: Intraoperative
Population: Per protocol analysis
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Experimental, IUD Insertion Group | Control, IUD Insertion Group
Number analyzed (Participants) | 108 | 107
score on a scale | 30 [0 to 86] | 38 [0 to 84]

ADVERSE EVENTS:
Time Frame: Adverse event data for each subject was assessed from time of consent to time of appointment discharge. On average this was 90 minutes.
Arm/Group | Experimental, IUD Insertion Group | Control, IUD Insertion Group
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/107
Other Adverse Events (participants affected / at risk) | 0/108 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02738203/Prot_SAP_000.pdf